CLINICAL TRIAL: NCT01675947
Title: Multi-Center, Randomized, Single Masked Phase 2 Study of Intravitreal Injections of Sirolimus in the Treatment of Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: Intravitreal Injections of Sirolimus in the Treatment of Geographic Atrophy
Acronym: Sirolimus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: On May 30, 2014, study injections were discontinued at the request of the DSMC. No further recruitment will occur.
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry); Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3368-12056; NCT01664208 (obsolete NCT alias)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — Sirolimus; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental): Monthly 20 μL (440 μg) intravitreal injection of sirolimus
  Interventions: Drug: Sirolimus
- Lidocaine (Sham Comparator): Monthly subconjunctival injection of 2% lidocaine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Sirolimus — Immunosuppressive agent. Blocks the T-lymphocyte activation and smooth muscle and endothelial cell proliferation that occurs in response to antigenic and cytokine (interleukin IL-2, IL-4 and IL-15) stimulation through either Ca2+-dependent or Ca2+-independent pathways. Sirolimus arrests cell cycle progression by direct interaction with two intracellular proteins (immunophilin FK binding protein 12 (FKBP-12) and the mammalian target of rapamycin (mTOR), a multifunctional serine-threonine kinase). In cells, sirolimus binds to FKBP-12, and the resulting sirolimus-FKBP-12 complex then binds to and inhibits mTOR.
  Other Names: Rapamycin, Rapamune
  Arms: Sirolimus
Drug: Lidocaine — Lidocaine 2%
  Other Names: Xylocaine; lignocaine
  Arms: Lidocaine

SUMMARY:
This study will seek to enroll 50 persons who have central or non-central geographic atrophy (GA) associated with age-related macular degeneration (AMD). GA in treated eye must be between 0.75 disk areas (DA) and 8 DA. Eligible participants will be randomly chosen to receive one of the following treatments in the study eye:

1. A 20 μL (440 μg) intravitreal (IVT) injection of sirolimus, or
2. A sham treatment (subconjunctival injection of lidocaine) Participants with two (2) eligible eyes will have one eye randomly assigned to receive intravitreal sirolimus and no sham in the fellow eye.

The first injection will begin at Day 0, which may occur on the date of screening/enrollment or up to two weeks following screening/enrollment visit, and every month thereafter. The visit schedule is as follows:

1. A clinical evaluation, including safety measures, will occur monthly.
2. Vision will be measured at the screening/enrollment visit and at 2, 3, 6, 9, 12, 18 and 24 months after the first injection has occurred.
3. Fundus autofluorescence will occur at screening/enrollment and at 2, 6, 12, 18 and 24 months after the first injection has occurred.
4. Fundus color photography and optical coherence tomography will occur at screening/enrollment and at 6, 12, 18 and 24 months after the first injection has occurred.

The primary goal is to evaluate whether the persons receiving the sirolimus injections show a slower worsening of geographic atrophy compared to the persons receiving the sham injections. A secondary goal is to evaluate the impact of sirolimus on vision compared to the sham.

NOTE: As of May 30, 2014, study injections were discontinued due to safety concerns. No further enrollments will occur and follow-up will continue on all active study participants on a quarterly basis. That is, on visits coinciding with 3 month intervals from date of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years of age or older. Prior participation in the Age-Related Eye Disease Study 2 (AREDS2) is not required.
* Participant must understand and sign the protocol's informed consent document.
* Participant must have central or non-central geographic atrophy (GA) in at least one eye. GA should be at least 0.75 disk areas (DA) in size but no more than 8 disk areas (DA); approximately 2.54 mm2 is 1 DA. GA is defined as one or more well-defined, usually more or less circular patches of partial or complete de-pigmentation of the retinal pigment epithelium (RPE), typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial de-pigmentation may still be classified as early GA.
* Participant must have a steady fixation in the study eye in the foveal or parafoveal area and media clear enough for good quality photographs.
* Participant must have visual acuity between 20/25 and 20/200 in the study eye.
* Female participants must be post-menopausal.
* Male participants with female partners capable of conceiving children will be required to use contraception during the study and for four months after their last sirolimus injection.

Exclusion Criteria:

* Participant is in another investigational study other than AREDS2 and actively receiving study therapy for geographic atrophy or choroidal neovascularization (CNV).
* Participant is unable to comply with study procedures or follow-up visits.
* Participant has evidence of ocular disease other than AMD in either eye that may confound the outcome of the study (e.g., glaucoma, diabetic retinopathy with 10 or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration, moderate/severe myopia).
* Participant has received treatment for AMD, such as macular laser, photodynamic therapy (PDT) or anti-vascular endothelial growth factor (anti-VEGF) therapy injection. Or the participant received an IVT injection of any agent (e.g., triamcinolone) other than an anti-VEGF agent within the last four months prior to study enrollment. Vitamin supplementation for AMD is not considered an exclusionary criterion.
* Participant has had a vitrectomy.
* Participant is expected to need ocular surgery during the course of the trial.
* Participant has undergone lens removal in the last three months or Yttrium Aluminium Garnet (YAG) laser capsulotomy within the last month.
* Participant is on chemotherapy.
* Participant is on immunosuppressive medication or is immunosuppressed.
* Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve.
* Participant with a history of malignancy that would compromise the 2-year study survival.
* Participant with a history of ocular herpes simplex virus (HSV).
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
* History of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years that could be worsened by immunosuppression. (The risk of immunosuppression must be determined by an oncology consultation prior to enrollment.)
* Ocular or periocular inflammation or infection in either eye.
* Presence of active or inactive toxoplasmosis in the study eye.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Rate of change in area of geographic atrophy | Every 6 months after enrollment for 2 years

SECONDARY OUTCOMES:
Change in best-corrected visual acuity | Every 6 months after enrollment for 2 years

OTHER OUTCOMES:
Number and severity of systemic and ocular toxicities, adverse events and infections | Monthly for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, MD, Study Chair — National Eye Institute (NEI)
Locations (13):
- United States (13):
  - Loma Linda University, Loma Linda, California
  - University of California, Davis, Sacramento, California
  - University of Florida HSC, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Elman Retina Group, Baltimore, Maryland
  - Vision Research Foundation, Grand Rapids, Michigan
  - Charlotte Eye Ear Nose & Throat Associates, Charlotte, North Carolina
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin